CLINICAL TRIAL: NCT03356002
Title: Evaluation of C-Scan System in Providing Structural Information and Detection of Polypoid Lesions in High Risk Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Check-Cap Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CL-SY-01-0094
Record Dates: First submitted 2017-11-20; First posted 2017-11-29 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: High Risk (Above Average) Subjects; Non Compliant Patients for Colo Rectal Cancer [CRC] Screening; Counterindicated Patients for Colonoscopy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: The colonoscopists will be blinded to the C-Scan system results and FIT results and the reviewers of C-Scan system results will be blinded to Fit and colonoscopy results
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High risk subjects (Active Comparator): Each subject will ingest the C-Scan System capsule within 30 days prior to colonoscopy. The results of the C-Scan review will be compared to the findings of colonoscopy.
  Subjects to be enrolled in this study are indicated and scheduled to undergo optical colonoscopy based on the following symptoms or by being classified as higher than average risk based on one or more of the following:
  c. Surveillance - Significant findings in previous optical colonoscopy d. Diagnostic - Polyps detected in virtual colonoscopy referred for polypectomy e. Diagnostic - Polyps detected in previous optical colonoscopy (community setting) referred for polypectomy f. Diagnostic - Positive FIT test g. Diagnostic - one or more of the typical symptoms:
  Interventions: Device: C-Scan System
- Average risk (Experimental): Each subject will ingest the C-Scan System capsule within 30 days prior to colonoscopy. The results of the C-Scan review will be compared to the findings of colonoscopy.
  Average risk based on their age and demographics referred for screening for polyps.
  Interventions: Device: C-Scan System

INTERVENTIONS:
Device: C-Scan System — Each subject will ingest the capsule within 30 days prior to colonoscopy. The results of the C-Scan review will be compared to the findings of colonoscopy.
  1. To establish the efficacy of C-Scan Capsule System and FIT in detecting patients with polypoid lesions ≥ 10mm, compared with Optical Colonoscopy
  2. To evaluate the safety of the C-Scan Capsule System procedure
  Other Names: Colon capsule

SUMMARY:
The purpose of this study is to establish the efficacy of Check-Cap's C-Scan System in providing structural information on colonic polypoid lesions and masses, as an adjacent tool to Feacal Immunochemical Test [FIT] in high risk subjects

DETAILED DESCRIPTION:
The subject will be invited to come to the clinic to sign the Informed Consent Form [ICF] and other related .

The subjects will be connected to the C-Scan Track and following system's activation the subject will be asked to ingest the C-Scan Capsule with some water and contrast media, in the presence of a physician.

Post ingestion, the subject will be discharged home with clear instructions on the procedure. The subject should avoid intensive physical exercise during procedure or any extreme activities. The subject should make an effort to stay at home or other familiar surroundings, and may continue daily activities such mobile/computer/Television use, shower, sleep or eat. Details on allowed and restricted activities are listed in app. 4 The subject will be required to ingest daily dose (3 X 15-17ml) of contrast media, to be consumed three times per day with normal diet. Also on a need based the subject would be provided with laxadine (5 mg tablets) to be ingested according to the doctor recommendation.

During capsule procedure the subjects will be contacted by phone several times daily by the site clinical study team (or by dedicated external trained medical personnel), to assure the subjects well-being and to monitor for any change or discomfort and for procedure progress. Subjects may be also monitored by the technical team (either at home or at the clinic), who may need to examine the system or inquire the subjects about the system visual/auditory indicators.

The subjects will be provided with a dedicated capsule collection kit, to assist the subjects in collecting the capsule. Subjects will be instructed to retrieve the capsule upon excretion.

Capsule procedure is completed upon capsule excretion or system vibro/auditory indication of 'End of Procedure'.

Once the procedure is completed, The C-Scan Capsule and C-Scan Track will be collected from the subject and returned to the sponsor's lab for preliminary analysis.

All subjects will be scheduled for optical colonoscopy to be performed within one month following capsule procedure.

C-Scan Procedure Analysis:

Several (3-6) licensed gastroenterologist physicians, will be trained with reviewing and analyzing C-Scan System scans, to serve as independent reviewers. Each case will be reviewed by 3 independant reviewers. The reviewing forum will be blinded to the FIT and colonoscopy results of the examined patients. Analysis will be performed on a per patient basis for the existence or non-existence of a finding that may be a polyp. This per patient finding will be compared with the FIT, and a colonoscopy will be performed for verification.

ELIGIBILITY:
Inclusion Criteria

* Male or female at the age of 40-80 years old
* Subject provided signed informed consent

Subjects to be enrolled in this study are indicated and scheduled to undergo optical colonoscopy based on the following symptoms or by being classified as higher than average risk based on one or more of the following:

Surveillance - Significant findings in previous optical colonoscopy Diagnostic - Polyps detected in virtual colonoscopy referred for polypectomy Diagnostic - Polyps detected in previous optical colonoscopy (community setting) referred for polypectomy Diagnostic - Positive FIT test

Diagnostic - one or more of the typical symptoms:

abdominal pain Change in bowel habits Anemia or overt bleeding in stool Significant weight loss

1st degree relatives of CRC subjects Alternatively average risk based on their age and demographics referred for screening for polyps.

Exclusion Criteria:

* Subjects with advanced cancer or other life threatening diseases or conditions
* Subject with known history of dysphagia or other swallowing disorders
* Subject with known history of GI disease or symptoms, such as: Crohn's disease, Colitis, Inflammatory Bowel Disease [IBD], Meckel's Diverticulum, Bowen Hernia, Mega Colon, fistulas or other strictures (doctors' discretion).
* Subject with known motility disorder or Chronic Constipation (less than 3 bowel movements/week)
* Subject with known delayed gastric emptying
* Subject with prior history of abdominal surgery that might cause bowel strictures leading to capsule retention, as determined by physician discretion
* Subject with any condition believed to have an increased risk for capsule retention such as intestinal tumors, radiation enteritis, and incomplete colonoscopies due to obstructions or NSAID enteropathy, as determined by physician discretion
* Subject with a cardiac pacemaker or other implanted electro medical device
* Subjects with known sensitivity to iodine, or with kidney failure
* Subjects with morbid obesity (BMI > 40)
* Subjects with belly / girth circumference > 125 cm
* Subject with any known condition which precludes compliance with study and/or device instructions
* Subject with known condition of drug abuse and/or alcoholism
* Subject who is unable to undergo colonoscopy or bowel preparation necessary for colonoscopy (based on previous attempts or self-declaration)
* Women who are either pregnant or nursing at the time of screening (to be verified by test in case of woman of child-bearing potential that do not practice medically acceptable methods of contraception)
* Concurrent participation in another clinical trial using any investigational drug or device

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2020-01-26 (Actual); Study Completion 2020-01-26 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of C-Scan Capsule System in detecting per segment polypoid lesions 10 mm and up as compared with Colonoscopy | One year
  Number of polyps detected by the capsule system in various segments of the colon as compared with the results indicated in the report of the follow-up colonoscopy

SECONDARY OUTCOMES:
Sensitivity and specificity of C-Scan Capsule System in detecting patients with polypoid lesions 6≤x≤9 mm, compared with Optical Colonoscopy | One year
  Number of polyp specificity of C-Scan Capsule System in detecting patients with polypoid lesions 6≤x≤9 mm detected by the capsule system in various segments of the colon as
Calculation of the score of the C-Scan system to generate a 3D model of the colon | One year
  Using the C-Scan View work station, the review will determine the score, on a scale of 1-10, the completeness of the colon model in each case. The average and Standard Deviation [SD] of all results will be calculated
Quantify the variance of the Interpretation of the data from the C-Scan System between the reviewers | One year
  Each case will be reviewed by 3 independent reviewers who are blinded to the results of the FIT and colonoscopy. Calculate the variance between the results of each reviewer

CONTACTS AND LOCATIONS:
Overall Officials: Boaz Shpigelman, Study Director — VP R&D
Locations (7):
- Israel (7):
  - Rambam Medical Center, Haifa, North
  - Haemek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Bnai-Zion Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Laniado Medical Center, Netanya
  - Tel Aviv Sorasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No
Preliminary results will be presented in the European Gastro Week Conference [UEGW] on October 2018